CLINICAL TRIAL: NCT06690437
Title: Observational Retrospective Multicentric Study for the Evaluation of the Clinical Performance and Safety Profile of the GALAXY FIXATION™ System and Orthofix Implantable Devices in Patients Who Have Needed Bone Stabilization or Bone Fixation for Fractures of the Long Bones, Vertically Stable Pelvic Fractures, or Vertically Unstable Pelvic Fractures As a Treatment Adjunct in Daily Practice: GALAXY Study
Brief Title: Observational Study for the Evaluation of the Clinical Performance and Safety Profile of the GALAXY FIXATION™ System and Orthofix Implantable Devices: GALAXY Study
Status: Active, not recruiting | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2204
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Fractures of the Long Bones; Vertically Stable Pelvic Fractures; Vertically Unstable Pelvic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Galaxy Fixation System and Orthofix implantable devices — It is planned to include 118 patients in 3 sites in Italy treated with GALAXY FIXATION™ System and Orthofix implantable devices for the following indications:
  * fractures of the long bones or;
  * Vertically stable pelvic fractures or vertically unstable pelvic fractures as a treatment adjunct Clinical data will be collected only from patients with a regular indication for GALAXY FIXATION™ System and Orthofix implantable devices as per IFUs (no off-label use will be included) and who underwent surgery performed with the specific devices.

SUMMARY:
The GALAXY FIXATIONTM System and Orthofix implantable devices study intends to evaluate the clinical performance and safety profile of the study medical/investigational devices in the standard clinical practice. The study will be conducted in three sites located in Italy considered reference sites for the treatment of adults and paediatric patients with fractures of the long bones, vertically stable pelvic fractures, or vertically unstable pelvic fractures as a treatment adjunct, where the usage of GALAXY FIXATION™ System and Orthofix implantable devices were part of the normal clinical practice. The participant investigators will retrospectively include a maximum of 118 patients in which GALAXY FIXATIONTM System and Orthofix implantable devices were used. No diagnostic or therapeutic intervention outside routine clinical practice will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. The patient directly or indirectly (through a respondent) expressed his willingness to participate in the Study by signing and dating informed consent.
2. Patient who had a regular indication for the following surgical intervention with the GALAXY FIXATION™ System and Orthofix implantable devices according to manufacturer's IFUs:

   * fractures of the long bones or;
   * Vertically stable pelvic fractures or vertically unstable pelvic fractures as a treatment adjunct.
3. Patients equal or older than 29 days.
4. Patients who had a regular indication for external fixation according to the investigator criteria.
5. Patients with clinical data registered in her/his medical records sufficient to assess the safety and efficacy endpoints of the study

Exclusion Criteria:

1. The patient is participating in other clinical studies or did he/she participate in the 3 months before signing the informed consent in other clinical studies.
2. The patient needed the application of or had already in-situ concomitant devices that couldn't be safely removed (except for permitted concomitant devices).
3. The patient was treated with more than one GALAXY FIXATION™ System or non Orthofix implantable devices.
4. Patient who had mental or physiological conditions who are unwilling or incapable of following postoperative care instructions.
5. Patient who had previous infections in the fracture area.
6. Patients who had malignancy in the fracture area.
7. Patients who had neuromuscular deficit or any other conditions that could influence the healing process.
8. Patients who had suspected or documented metal sensitivity reactions as it could result in a treatment failure in the intended population

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is planned to include 118 patients in 3 sites in Italy treated with GALAXY FIXATION™ System and Orthofix implantable devices for the following indications:
  * fractures of the long bones or;
  * Vertically stable pelvic fractures or vertically unstable pelvic fractures as a treatment adjunct Clinical data will be collected only from patients with a regular indication for GALAXY FIXATION™ System and Orthofix implantable devices as per IFUs (no off-label use will be included) and who underwent surgery performed with the specific devices.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The clinical performance of GALAXY FIXATION™ System and Orthofix implantable devices. | average of 2 months
  It will be assessed by the percentage of patients in which GALAXY FIXATION™ System and Orthofix implantable devices have guaranteed the maintenance of reduction in temporary stabilization and the achievement of bone union in definitive fixation until the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alessando Casiraghi, MD, Principal Investigator — Spedali Civili di Brescia
Locations (3):
- Italy (3):
  - Spedali Civili di Brescia, Brescia
  - Ospedale Niguarda Ca' Granda di Milano, Milan
  - Ospedale di Vicenza, Vicenza